CLINICAL TRIAL: NCT03595878
Title: Randomized Trial of Parotid Sparing Whole Brain Radiation
Brief Title: Trial of Parotid Sparing Whole Brain Radiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); University of Michigan (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LCCC 1802
Record Dates: First submitted 2018-05-18; First posted 2018-07-23 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2023-03

CONDITIONS: Xerostomia
Keywords: Whole Brain Radiation
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Randomized Arm - Control Group (Active Comparator): Patients randomized to this group will receive standard WBRT.
  Interventions: Radiation: Standard WBRT
- Randomized Arm - Intervention Group (Experimental): Patients randomized to this group will receive parotid sparing WBRT.
  Interventions: Radiation: Parotid sparing WBRT
- Observational Arm (No Intervention): Patients enrolled in this arm will be treated per their treating physician's choice.

INTERVENTIONS:
Radiation: Parotid sparing WBRT — Whole Brain Radiation Therapy with avoidance of the parotid glands
  Arms: Randomized Arm - Intervention Group
Radiation: Standard WBRT — Standard Whole Brain Radiation Therapy
  Arms: Randomized Arm - Control Group

SUMMARY:
The purpose of this study is to evaluate the efficacy of parotid sparing in reducing measurable xerostomia (dry mouth) in patients undergoing whole brain radiotherapy. This is primarily a two-arm, single-blind, randomized study of parotid sparing whole brain radiation therapy (WBRT), with a third observational arm of patients who were identified after radiation had already started or who refused randomization but were willing to be followed for quality of life assessment. Qualifying patients who are interested in participating in the trial will be asked to complete an anonymous screening baseline xerostomia questionnaire. If their raw score on this questionnaire meets eligibility criteria, they will be offered enrollment on the study. Patients identified prior to radiation start will be offered enrollment into the interventional randomization arm, with the observation arm offered to those who refuse randomization. Patients identified after radiation has already started, but within 5 days of the first day of radiation, will be offered enrollment into the observational arm. Questionnaires completed by patients who consent to the trial will be assigned patient information (de-anonymized) and serve as their baseline quality of life data. After baseline assessment, subjects will be asked to complete the same questionnaire again at the end of treatment, as well as two weeks, one month, three months, and six months after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be treated with WBRT using 3-dimensional conformal RT in 10-15 fractions to a total dose of 30-35 Gy for any diagnosis other than elective treatment of potentially subclinical intracranial disease.
* No prior radiation that would have exposed the parotids to a significant level of radiation (estimated >10 Gy mean parotid dose). Patients receiving prior stereotactic radiosurgery for brain metastasis are eligible for inclusion in this trial as this form of radiation is highly conformal and exposes the parotids to minimal (estimated <1 Gy) radiation.

  * Patients enrolling on the observational arm may have started their current course of whole brain radiation therapy within 5 days prior to completing the baseline screening questionnaire and consenting to study.
* Greater than or equal to 18 years of age (no upper age limit).
* Raw xerostomia score < 40 / 80 on the initial screening xerostomia questionnaire. This is calculated by adding up the values from questions 1-8.
* Initial xerostomia questionnaire and informed consent obtained within the required time frame (≤ 30 days before RT start for interventional arm; ≤ 5 days after RT start for observational arm).

Exclusion Criteria:

* Patients receiving WBRT without the use of a CT- or MRI-based planning simulation.
* Patients receiving WBRT with the use of intensity-modulated radiation therapy.
* Patient receiving WBRT as elective treatment of potentially subclinical intracranial disease (e.g., WBRT for prophylactic cranial irradiation of small cell lung cancer).
* Patients physically unable to communicate by paper or phone to complete the study survey.
* Prisoners.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colette Shen, Principal Investigator — University of North Carolina at Chapel Hill, Department of Radiation Oncology
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina
  - Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 05/09/2018 through 02/03/2021 at 3 cancer centers in the United States.
Pre-assignment Details: Sixty subjects were included in the study: 56 subjects were randomized into 2 groups: Group A (29 subjects) and Group B (27 subjects), and 4 subjects who started therapy according to physician choice, were included in Group C.
Groups:
- Arm A: Randomized Control Group: Subjects received standard whole-brain radiation therapy
- Arm B: Randomized Intervention Group: Subjects received standard whole-brain radiation therapy with avoidance of the parotid glands.
- Arm C: Observational Arm: Subjects enrolled in this arm per their physician's choice, received standard whole-brain radiation therapy.
Period: Overall Study
Arm/Group | Arm A: Randomized Control Group | Arm B: Randomized Intervention Group | Arm C: Observational Arm
Started | 29 | 27 | 4
Completed | 25 | 25 | 2
Not Completed | 4 | 2 | 2
Not completed — Death | 2 | 1 | 0
Not completed — Disease progression | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Subjects undergoing whole brain radiotherapy enrolled in the study and assessed per study criteria.
Groups:
- Arm A:RandomizedControl Group: Subjects received standard whole-brain radiation therapy
- Arm B:RandomizedIntervention Group: Subjects received standard whole-brain radiation therapy with avoidance of the parotid glands.
- Arm C:Observational Arm: Subjects enrolled in this arm per their physician's choice, received standard whole-brain radiation therapy.
- Total: Total of all reporting groups
Arm/Group | Arm A:RandomizedControl Group | Arm B:RandomizedIntervention Group | Arm C:Observational Arm | Total
Number analyzed (Participants) | 29 | 27 | 4 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 15 | 4 | 39
  >=65 years | 9 | 12 | 0 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 1 | 35
  Male | 12 | 10 | 3 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 25 | 4 | 58
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 1 | 7
  White | 27 | 22 | 3 | 52
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 27 | 4 | 60

OUTCOME MEASURES:

1. Primary Outcome: Xerostomia One Month After Completion of Treatment
Description: Between baseline and 1 month after the treatment xerostomia symptoms were assessed, in 2 randomized groups namely Arm A and Arm B.
  Xerostomia symptoms were assessed using the patient-reported study xerostomia questionnaire. The questionnaire includes 8 questions, and each question score changes between 0 to 10. The increasing value represents worse xerostomia symptoms. No xerostomia symptom= 0 and highest xerostomia symptom=10. The total score will be on a scale from 0-80 (8 categories with a maximum score of 10).
  Changes in xerostomia symptoms in each arm were tabulated. Positive values represent increased xerostomia symptoms and negative values represent decreasing xerostomia symptoms and no difference is no change.
Time Frame: Up to 45 days
Population: Subjects were randomized in 2 randomized groups namely Arm A and Arm B, completed the treatment, and responded to the quality-of-life questionnaire, both at baseline and after 1 month after completion of treatment. Arm C was not included since Arm C is not a randomized arm.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Arm - Control Group: Subjects randomized to this group receive Standard Whole Brain Radiation Therapy (WBRT).
- Randomized Arm - Intervention Group: Subjects randomized to this group will receive parotid-sparing Whole Brain Radiation Therapy (WBRT), with avoidance of the parotid glands.
Arm/Group | Randomized Arm - Control Group | Randomized Arm - Intervention Group
Number analyzed (Participants) | 15 | 18
Participants
  Improved: Decreased xerostomia symptoms | 5 | 7
  No Change in xerostomia symptoms | 1 | 6
  Worsened: Increased xerostomia symptoms | 9 | 5

2. Secondary Outcome: Freedom From Relapse
Description: The number of subjects with marginal cervical spine relapse in each randomization arm.
Time Frame: Up to 6 months
Population: The subjects completed the treatment and were assessed for the occurrence of marginal relapse.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A Randomized Arm - Control Group: Patients randomized to this group receive standard Standard Whole Brain Radiation Therapy (WBRT).
- Arm B Randomized Arm - Intervention Group: Patients randomized to this group will receive parotid-sparing Whole Brain Radiation Therapy (WBRT), with avoidance of the parotid glands.
- Arm C : Not- Randomized Arm Observational Arm: Patients enrolled in this arm were not randomized, they are enrolled per their treating physician's choice.
Arm/Group | Arm A Randomized Arm - Control Group | Arm B Randomized Arm - Intervention Group | Arm C : Not- Randomized Arm Observational Arm
Number analyzed (Participants) | 15 | 14 | 1
Participants
  Number of subject with marginal relapse | 0 | 0 | 0
  Number of subject without marginal relapse | 15 | 14 | 1

3. Secondary Outcome: Xerostomia Based on Radiotherapy Treatment Fields- One Month After the Treatment
Description: Between baseline and 1 month after the treatment xerostomia symptoms were assessed and tabulated based on the whole brain radiotherapy (WBRT) technique. The Standard WBRT Group includes both randomized (Group A) and non-randomized (Group C) subjects who received WBRT. The Parotid Sparing WBRT Group includes subjects who were randomized and received Parotid Sparing WBRT (Group B). Xerostomia symptoms were assessed using the patient-reported study xerostomia questionnaire. The questionnaire includes 8 questions, and each question score changes between 0 to 10. The increasing value represents worse xerostomia symptoms. No xerostomia symptom= 0 and highest xerostomia symptom=10. The total score will be on a scale from 0-80 (8 categories with a maximum score of 10). Changes were tabulated as: Positive values represent worsened xerostomia symptoms, and both negative values and no change values represent did not worsen.
Time Frame: Up to 45 days
Population: Subjects completed the treatment and responded to the quality-of-life questionnaire both at baseline and one month after the treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Whole Brain Radiation Therapy- Arm A: The Standard WBRT Group includes randomized subjects (Group A)
- Parotid Sparing Whole Brain Radiotherapy: Subjects received parotid-sparing whole-brain radiotherapy (Arm B).
- Standard Whole Brain Radiation Therapy- Arm C: The Standard WBRT Group includes non-randomized (Group C) subjects who received WBRT.
Arm/Group | Standard Whole Brain Radiation Therapy- Arm A | Parotid Sparing Whole Brain Radiotherapy | Standard Whole Brain Radiation Therapy- Arm C
Number analyzed (Participants) | 15 | 18 | 1
Participants
  Xerostomia Worsened | 9 | 5 | 0
  Xerostomia did not worsen | 6 | 13 | 1

ADVERSE EVENTS:
Time Frame: Not available. The protocol does not require adverse event assessment.
Description: The protocol does not require adverse event assessment. Adverse Event Data was not collected.
Groups:
- Arm A:Randomized Control Group: Subjects receive standard whole-brain radiation therapy
- Arm B:Randomized Intervention Group: Subjects received standard whole-brain radiation therapy with avoidance of the parotid glands.
- Arm C: Observational Arm: Subjects enrolled in this arm per their physician's choice, receive standard whole-brain radiation therapy.
Arm/Group | Arm A:Randomized Control Group | Arm B:Randomized Intervention Group | Arm C: Observational Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators' joint publication is required.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT03595878/Prot_SAP_000.pdf